CLINICAL TRIAL: NCT05471635
Title: Determinants of COVID-19 Vaccination Worldwide: WORLDCOV, a Retrospective Observational Study
Brief Title: Variables Influencing Anti-COVID-19 Vaccinations Around the World: an Analysis Conducted on Aggregated Data Sourced From Institutional Databases to Understand Whether and How Different Variables Could Affect the Vaccine Coverage (WORLDCOV: Worldwide Determinants of COVID-19 Vaccination)
Acronym: WORLDCOV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Alberto Peano (Other)
Responsible Party: Sponsor-Investigator, Alberto Peano, MD, Resident doctor in Public Health, Department of Public Health Sciences and Pediatrics, University of Turin, Italy
Organization: University of Turin, Italy (Other)
Other Study IDs: GP0012022
Record Dates: First submitted 2022-07-20; First posted 2022-07-25 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: COVID-19 Vaccines
MeSH Terms: interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Countries worldwide: Every country in the world for which vaccination data were available and variables of interest were accessible.
  Interventions: Biological: COVID-19 Vaccine

INTERVENTIONS:
Biological: COVID-19 Vaccine — All COVID-19 vaccines approved by national or international regulatory agency, despite the vaccine technology, manufacturer, and regulatory agency that granted marketing authorization.

SUMMARY:
Vaccination coverage against COVID-19 differs widely between countries: in order to address this public health issue, this observational study seeks to understand whether there are any determinants/predictors. In order to highlight the presence of determinants and their strength in influencing vaccination coverage, all possible socio-demographic, economic, cultural, infrastructural and political variables considered capable of modifying such coverage were selected and analysed.

DETAILED DESCRIPTION:
The COVID-19 pandemic has had major health, economic and social implications, bringing with it a large number of deaths worldwide. While the lethality rate could not be considered high, the fact that the contagiousness was high resulted in a considerable number of deaths. As a result, the COVID-19 pandemic has become a sudden, huge and urgent public health problem.

Initially faced with a new and unknown etiopathological entity, different countries adopted different policies that proved more or less effective in containing the COVID-19 contagion. While social and hygienic restrictive measures (i.e. so-called social distancing, curfews, use of masks and hand hygiene) initially had a positive impact on reducing infections, for the most part they proved to be ephemeral measures. These actions were short-lived because they were not sustainable over time due to the damage they implied with regard to mental health, besides the low adherence of the population. A relaxation of these restrictive measures has always led to an increase in the spread of the COVID-19 pandemic, with a resurgence of hospital admissions, an ever-increasing occupancy of intensive care beds and a subsequent increase in the number of deaths.

Since the beginning of the COVID-19 pandemic, scientific research has been working to enable the identification of the SARS-CoV-2 viral genome and possible target proteins for treatment. Due to years of vaccine research and the launch of Access to COVID-19 Tools (ACT)-Accelerator partnership, a rapid development of several candidate vaccines based on different vaccine technologies and thus to their rapid clinical testing were possible.

Thanks also to the regulatory agencies' solicitude, in certain Countries (e.g. Israel, the UK, the US and the EU) the COVID-19 vaccination campaign started at the end of 2020 and extended worldwide during 2021 (with the exception of Eritrea and the Democratic Republic of Korea).

Through purchasing agreements with individual vaccine manufacturers, governments (or supranational institutions, e.g. the EU) secured the supply of the necessary doses. However, this entailed a division of the world's population depending on the negotiating power of the country of residence and, therefore, its economic strength. COVAX is one of the three pillars of the ACT-Accelerator programme: dedicated to vaccines, the purpose of COVAX is to accelerate the development and manufacture of COVID-19 vaccines, ensuring fair and equitable access for every country in the world.

In a globalised world, guaranteeing everyone the right to health is mandatory from a moral as well as an economic and global health point of view: everyone gains if the poorest improve their condition (think infectious diseases). In a globalised world, it is necessary to 'globalise' health and not only the economy: this study aims to understand where governments, supranational institutions and non-governmental organisations can act more incisively to combat the COVID-19 pandemic with the weapon the vaccine represents.

On this basis, the investigators decided to examine whether certain variables could be determinants of vaccination coverage for COVID-19. Two outcomes were identified as indicators of vaccination coverage: the proportion of the population vaccinated with at least one dose and the ratio of administered doses to the population. These data were obtained from the COVID-19 dataset by Our World In Data as of 15th June for each country. If data was not available on that date, the most recent available data was used looking retrospectively. In order to analyze whether and which were determinants of vaccination coverage, several variables are accounted: socio-demographic variables: total population, population density, median age, GINI Index; economic variables: GDP per capita; health variables: COVID-19-specific mortality, type of health system (public or private), health personnel (Physicians /1000 population, Nurses and midwives personnel/1000 population); cultural variables (literacy rate, Greenberg Index, presence of a predominant religion), infrastructural variables (density of road network, access to electricity) and political variables (civil liberties, political stability and absence of violence/terrorism). Data for the aforementioned variables were extracted from institutional databases/ datasets: World Bank, Our World In Data, World Religion Database and The World Factbook. For Greenberg Index, as proxy of Cultural Diversity Index, the data were from Gören (2018), taking the 2020 figure for each country, or the most recent available figure if the 2020 figure is not available.

Statistical analyses will be conducted including all countries in the world taken individually, for which vaccination data are available as of 15 June 2022. In addition, analyses will also be conducted for outcomes adjusted for vaccine doses delivered (in each country). The data for this correction factor were obtained from the UNICEF database on 21th June 2022.

Statistical analyses by subgroups will also be implemented, stratifying by World Bank country classification by income level: High, Upper-middle, Lower-middle, Low.

ELIGIBILITY:
Inclusion Criteria:

* All countries (independent or not) in the world

Exclusion Criteria:

* No data available on vaccination coverage and dose administered population ratio
* Substantial lack of data

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All countries worldwide, if not excluded in reason of Exclusion Criteria
Sampling Method: Non-Probability Sample
Enrollment: 205 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-07-20 (Estimated); Study Completion 2022-07-20 (Estimated)

PRIMARY OUTCOMES:
Vaccination coverage | 15th June 2022 for each country, independently from the beginning date of the COVID-19 vaccination campaign
  Proportion of the population vaccinated with at least one dose
Total doses administered per 100 residents | 15th June 2022 for each country, independently from the beginning date of the COVID-19 vaccination campaign
  Doses of vaccine administered per 100 population in each country, that is the ratio of administered doses to the population

CONTACTS AND LOCATIONS:
Overall Officials: Maria M Gianino, Prof., Study Director — University of Turin, Department of Public Health Sciences and Pediatrics; Alberto Peano, Dr., Principal Investigator — Department of Public Health Sciences and Pediatrics, University of Turin; Gianfranco Politano, PhD, Principal Investigator — Department of Control and Computer Engineering, Polytechnic University of Turin
Locations (1):
- University of Turin, Turin, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Peano A, Politano G, Gianino MM. Determinants of COVID-19 vaccination worldwide: WORLDCOV, a retrospective observational study. Front Public Health. 2023 Aug 31;11:1128612. doi: 10.3389/fpubh.2023.1128612. eCollection 2023. PMID 37719735